CLINICAL TRIAL: NCT04321382
Title: Subjective Perception of Ocular Prosthesis Wear
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s61570
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Anophthalmos, Unilateral; Prosthesis User
MeSH Terms: conditions — Anophthalmos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The loss of an eye, whether congenital or acquired, is a severe psychological trauma with negative impact on the quality of life of the patient. While rehabilitation with a customized ocular prosthesis anatomically restores the facial appearance, the final outcome is largely determined by the subjective satisfaction of the patient. By investigating the level of subjective perception, the quality of care can be improved.

ELIGIBILITY:
Inclusion Criteria:

* acquired anophthalmia
* Informed consent
* ocular prosthesis wear for minimum of 2 years

Exclusion Criteria:

* congenital anophthalmia
* microphthalmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unilateral anophthalmic patients wearing an ocular prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Quality of care | 1 hour
  disease specific score

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruiters S, De Jong S, Mombaerts I. Measuring quality of care and life in patients with an ocular prosthesis. Graefes Arch Clin Exp Ophthalmol. 2021 Jul;259(7):2017-2025. doi: 10.1007/s00417-021-05088-1. Epub 2021 Feb 6. PMID 33547966